CLINICAL TRIAL: NCT00028574
Title: A Phase III Randomized, Double-Blind, Placebo-Controlled Trial of Gabapentin in the Management of Hot Flashes in Men
Brief Title: Gabapentin in Treating Hot Flashes in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NCCTG-N00CB; NCCTG-N00CB; NCI-P01-0199; CDR0000069107 (Registry Identifier: NCI Physician Data Query); NCI-2012-02435 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Hot Flashes; Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; hot flashes
MeSH Terms: conditions — Hot Flashes; Prostatic Neoplasms | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Gabapentin (28 days) (Active Comparator): Oral Gabapentin 300 mg days 1-28
  Interventions: Drug: gabapentin
- Gabapentin (7, 21) (Active Comparator): Oral Gabapentin 300 mg once daily on days 1-7 days and twice daily days 8-28
  Interventions: Drug: gabapentin
- Gabapentin (7, 7, 14) (Active Comparator): Oral Gabapentin 300 mg once daily on days 1-7, twice daily on days 8-14 and three times daily on days 15-28
  Interventions: Drug: gabapentin
- Placebo (Placebo Comparator): Oral Placebo 300 mg on one of the following schedules:
  * once daily on days 1-28
  * once daily on days 1-7, twice daily on days 8-28
  * once daily on days 1-7, twice daily on days 8-14 and three times daily on days 15-28
  Interventions: Other: placebo

INTERVENTIONS:
Drug: gabapentin
  Arms: Gabapentin (28 days); Gabapentin (7, 21); Gabapentin (7, 7, 14)
Other: placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Gabapentin may be effective in relieving hot flashes in men who have prostate cancer. It is not yet known which regimen of gabapentin is most effective in treating hot flashes.

PURPOSE: Randomized phase III trial to compare different regimens of gabapentin in treating men who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of gabapentin in managing hot flashes in men with prostate cancer.
* Determine the response of patients to this drug.
* Determine the toxicity of this drug in these patients.
* Determine the quality of life of patients treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to the number of hot flashes per day (2-3 vs 4-9 vs 10 or more) and duration of hot flash symptoms (less than 9 months vs 9 months or more). Patients are randomized to one of four treatment arms.

All patients are observed for 7 days prior to drug administration in order to collect baseline hot flash information.

* Arm I: Patients receive oral gabapentin once daily on days 1-28.
* Arm II: Patients receive oral gabapentin once daily on days 1-7 and twice daily on days 8-28.
* Arm III: Patients receive oral gabapentin once daily on days 1-7, twice daily on days 8-14, and three times daily on days 15-28.
* Arm IV: Patients receive oral placebo on one of three schedules corresponding to arms I-III.

Patients in all arms may continue therapy with gabapentin for an additional 8 weeks.

Quality of life is assessed at baseline, day 28, and at the end of the additional 8 weeks.

Patients are followed at 6, 12, and 24 months.

PROJECTED ACCRUAL: A total of 220 patients (55 per treatment arm) will be accrued for this study within 1 year.

ELIGIBILITY:
Required characteristics:

1. Men with a history of prostate cancer who have received or are receiving androgen ablation therapy.
2. Must be on a stable dose of hormone therapy for the past 4 weeks and must not be planning on discontinuing hormone therapy throughout the duration of the randomized phase (5 weeks).
3. Presence of hot flashes for ≥1 month prior to study entry.
4. Bothersome hot flashes (defined by their occurrence ≥14 times per week and of sufficient severity to make the patient desire therapeutic intervention).
5. Life expectancy ≥ 6 months.
6. ECOG Performance Status (PS) 0 or 1.
7. ≥18 years of age

Contraindications:

1. History of renal insufficiency (defined as a creatinine ≥1.5 x UNL in the last two years).
2. Any of the following current (≤ 4 weeks) or planned therapies:

   * Antineoplastic chemotherapy
   * Androgens
   * Estrogens
   * Progestational agents
3. History of allergic or other adverse reaction to gabapentin.
4. Prior use of gabapentin.
5. Antidepressants (use is allowed if patient has been on a stable dose for ≥1 month and does not plan to modify this treatment during the next 5 weeks).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2001-12; Primary Completion 2006-12 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Hot flash reduction by diary scores at 4 weeks | 5 weeks from study entry

SECONDARY OUTCOMES:
Toxicity by questionnaires at 4 weeks | 5 weeks from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, MD, Study Chair — Mayo Clinic
Locations (170):
- United States (170):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Howard University Cancer Center at Howard University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Cancer Research Center of Hawaii, Honolula, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Leeward Radiation Oncology Center, ‘Ewa Beach, Hawaii
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Albert Lea Cancer Center at Albert Lea Medical Center, Albert Lea, Minnesota
  - Alexandria, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fergus Falls, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Sartell, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Clinic of Dr. Judy L. Schmidt, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Loprinzi CL, Dueck AC, Khoyratty BS, Barton DL, Jafar S, Rowland KM Jr, Atherton PJ, Marsa GW, Knutson WH, Bearden JD 3rd, Kottschade L, Fitch TR. A phase III randomized, double-blind, placebo-controlled trial of gabapentin in the management of hot flashes in men (N00CB). Ann Oncol. 2009 Mar;20(3):542-9. doi: 10.1093/annonc/mdn644. Epub 2009 Jan 6. PMID 19129205
- [Result] Moraska AR, Atherton PJ, Szydlo DW, Barton DL, Stella PJ, Rowland KM Jr, Schaefer PL, Krook J, Bearden JD, Loprinzi CL. Gabapentin for the management of hot flashes in prostate cancer survivors: a longitudinal continuation Study-NCCTG Trial N00CB. J Support Oncol. 2010 May-Jun;8(3):128-32. PMID 20552926